CLINICAL TRIAL: NCT02894632
Title: MR Compatible Accelerometer for Respiratory MOTion Measurement
Acronym: MARMOT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2012-A00874-39
Record Dates: First submitted 2016-08-24; First posted 2016-09-09 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-09

CONDITIONS: Heart Disease
Keywords: MRI; Motion; Respiratory movement; Artifacts correction
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Healthy volunteers (Experimental): Volunteers without cardiac, hepatic or renal pathology
  Interventions: Device: MRI compatible motion sensor (MARMOT)

INTERVENTIONS:
Device: MRI compatible motion sensor (MARMOT) — MRI with motion control (several motion sensors placed on the volunteer's body)

SUMMARY:
A novel magnetic resonance (MR) compatible accelerometer for respiratory motion sensing (MARMOT) has been developed as a surrogate of the vendors' pneumatic belts. The aim is to model and correct respiratory motion for free-breathing thoracic-abdominal MR imaging and to simplify patient installation.

DETAILED DESCRIPTION:
Respiratory motion is a serious problem in the acquisition of high-quality thoracic/abdominal magnetic resonance (MR) images. Various methods have been proposed to compensate the motion-induced artefacts, including breathholding, respiratory gating and model-driven motion correction.

Breath-holding is the simplest among the three. However this conventional clinical method induces various problem, including inefficient use of scanners, inconsistent organ position between each breath-hold, imaging an altered physiological status and patient inconvenience especially for those who suffer from respiration difficulties. Free-breathing MR acquisition has therefore become of great clinical interest recently.

The investigators intend to examine the efficacy of the MARMOT sensors for:

* modelling and predicting the respiratory motions in abdominal scans,
* correcting for the respiratory motion in a cardiac cine scan, via a reconstruction-based method.

ELIGIBILITY:
Inclusion Criteria:

* To not have cardiac, hepatic or renal pathology
* To be more than 18
* To be enrolled in a social security plan
* To have signed an informed consent
* To have preliminary medical examination

Exclusion Criteria:

* Contraindication: implantable devices (pacemakers, defibrillators, cochlear implants, etc.), metallic foreign bodies
* Impossibility to undergo MRI : claustrophobia, morbid obesity
* Pregnancy or risk of pregnancy
* Patient under a measure of legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-07; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Respiratory movement using respiratory belts | four months
  Respiratory belts, which are usually used in MRI to monitor respiratory movements and brath-holding, are placed around the volunteer's body (on the abdominal and on the thoracic level).
  They give the average displacement (in mm) across time generated by the respiratory movement.
Respiratory movement using MARMOT sensors | four months
  MARMOT sensors are placed on the volunteer's body (4 sensors placed on the thorax or on the abdomen).
  MARMOT sensors give 2 measures : acceleration generated by the respiratory movement (in mm/s²) in 3 directions and rotation generated by the respiratory movement (angle in °/s) in 3 directions.
Respiratory movement using real-time MR images | four months
  Motion measurement (in mm) directly on the MR images (using real-time MR imaging)

SECONDARY OUTCOMES:
Subjective quality (marks between 1 (the best) and 3 (the worst) of the reconstructed MR images) | four months
  Comparing the quality of the reconstructed cardiac cine images obtained with the cine-GRICS algorithm using:
  * the pneumatic belts alone
  * all MARMOT signals
  * signals from only one MARMOT sensor.
  Three cardiologists are shown with the motion-compensated cine movies obtained using these three sensor configurations. The movies are presented in random ordering on the screen so that the clinicians are blind to the sensor configuration. They are then asked to rank them by overall image quality (1=best, 2=second best, 3=worst). Equal quality ranking is allowed in this procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Bonnemains, Dr, Principal Investigator — Inserm - U947
Locations (1):
- Centre Hospitalier Régional Universitaire de Nancy Brabois, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No